CLINICAL TRIAL: NCT07072455
Title: Sensory Profile of People With High Intellectual Potential
Brief Title: Sensory Profile of People With High Intellectual Potential (HIP)
Acronym: HPIsens
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Aude Paquet, Psychomotor Therapist, Doctor in Psychology, Centre Hospitalier Esquirol
Other Study IDs: 2024-A02488-39
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: High Intellectual Potential
Keywords: High Intellectual Potential; Sensory Profile; Coping Strategies; Anxiety; Sensory Processing; Autistic traits
MeSH Terms: conditions — Anxiety Disorders | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Intellectual Potential: Subjects with a High Intellectual Potential : Cognitive assessment using the Wechsler Adult Intelligence Scale (WAIS-III or WAIS-IV) scale or Wechsler Intelligence Scale for Children (WISC-VI or WISC-V) scale by a psychologist.
  Intelligence Quotient (IQ) ≥ 130, in the case of a homogeneous cognitive profile, or General Aptitude Index (GAI) ≥ 130 [124-134], in the case of a heterogeneous cognitive profile
  Interventions: Other: Scales; Other: High Intellectual Potential Scale
- Control: Subjects whitout High Intellectual Potential
  Interventions: Other: Scales

INTERVENTIONS:
Other: Scales — This observational study consists of data collection using a structured questionnaire based on an e-CRF, distributed by e-mail.
  Four questionnaires were administered : the Revised Ritvo Autism and Asperger Diagnostic Scale (RAADS-R-Fr), the Adolescent/Adult Sensory Profile (AASP), the Coping Inventory for Stressful Situations (CISS) and the State-Trait Anxiety Inventory (STAI-Y).
  Socio-demographic and treatments were collected.
Other: High Intellectual Potential Scale — For participants with High Intellectual Potential, the total Intelligence Quotient (IQ) or General Ability Index (GAI), along with the index scores from the Wechsler scales (Verbal Comprehension Index, Perceptual Reasoning Index, Working Memory Index, and Processing Speed Index), will be extracted from the cognitive assessment previously completed by the participant prior to study enrollment.
  Groups: High Intellectual Potential

SUMMARY:
This is a prospective observational psychology study on a non-clinical population, involving the use of questionnaires (non-interventional research).

This study involves the collection of data associated with High Intellectual Potential characteristics, sensory profile, and includes clinical measures such as anxiety anxiety, autistic traits and coping in High Intellectual Potential and control participants.

ELIGIBILITY:
Inclusion Criteria:

* High Intellectual Potential:
* Participants with a High Intellectual Potential : Cognitive assessment using the WAIS or WISC-V scale by a psychologist; Intelligence Quotient (IQ) ≥ 130, in the case of a homogeneous cognitive profile, or General Aptitude Index (GAI) > 130 [124-134], in the case of a heterogeneous cognitive profile
* Gender and Age: Male or female, aged 18 to 65
* Consent: Free, informed, and written consent (e-CRF)
* Control :
* Gender and Age: Male or female, aged 18 to 65
* Consent: Free, informed, and written consent (e-CRF)

Exclusion Criteria:

* High Intellectual Potential:
* History or declared psychiatric disorder (characterized depressive episode, personality disorder, addiction, eating disorder, bipolar disorder, obsessive-compulsive disorder)
* Neurodevelopmental disorders (autism spectrum disorder, attention deficit and hyperactivity disorder , developmental coordination disorder)
* Sensory disability
* Subjects under guardianship or curatorship
* Pregnant or breast-feeding women
* Control :
* Presence of High Intellectual Potential known
* Presence of intellectual development disorder
* History or declared psychiatric disorder (characterized depressive episode, personality disorder, addiction, eating disorder, bipolar disorder, obsessive-compulsive disorder)
* Neurodevelopmental disorders (autism spectrum disorder, attention deficit and hyperactivity disorder , developmental coordination disorder)
* Sensory disability
* Subjects under guardianship or curatorship
* Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with High Intellectual Potential will be recruited on a voluntary basis :
  * in the offices of private psychologists, on the psychologist's recommendation or by posting in waiting rooms
  * through communication on social networks Subjects control will be recruited on a voluntary basis from the personal and professional environment of the people involved in this study and through communication on social networks.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Sensory profile from the Adolescent and Adult Sensory Profile according to each group. | At enrollment
  Sensory profile scores is obtained using the self-report questionnaire Adolescent and Adult Sensory Profile (AASP) after the participant has been included in the study. Subscores for sensory sensitivity, low registration, sensation seeking, and sensation avoidance are collected. For each subscore, the minimum and maximum values range from 15 to 75. A high score indicates high sensory sensitivity.

SECONDARY OUTCOMES:
Sensory profile from the Adolescent and Adult Sensory Profile according to the cognitive profile of the High Intellectual Potential group. | At enrollment
  Sensory profile scores will be obtained using the Adolescent and Adult Sensory Profile (AASP) scale during an individual interview after the participant has been included in the study. Subscores for sensory sensitivity, low registration, sensation seeking, and sensation avoidance will be collected. For each subscore, the minimum and maximum values range from 15 to 75. A high score indicates high sensory sensitivity.
Scores for anxiety from the State and Trait Anxiety Inventory according to each group | At enrollment
  Anxiety scores will be obtained using the State and Trait Anxiety Inventory (STAI-Y) scale during an individual interview after the participant has been included in the study. Subscores for State Anxiety and Trait Anxiety will be collected. For each subscore, the minimum and maximum values range from 20 to 80. A high score indicates high anxiety
Scores for task coping drawn from the Coping Inventory for Stressful Situations according to each group | At enrollment
  Coping scores will be obtained using the Coping Inventory for Stressful Situations (CISS) scale during an individual interview after the participant has been included in the study. The task-oriented coping subscore, emotion subscore, avoidance subscore, distraction subscore, and social diversion subscore will be collected. The minimum and maximum values range from 16 to 90. A high score indicates high oriented coping.
Description of the frequency of autistic traits for each group | At enrollment
  The frequency of autistic traits will be obtained using the Revised Ritvo Autism and Asperger Diagnostic Scale (RAADS-R-Fr) during an individual interview after the participant has been included in the study. The minimum and maximum values range from 0 to 240. The generally accepted threshold for significant autistic traits is 70. A high score indicate high autistic traits.

CONTACTS AND LOCATIONS:
Locations (1):
- Esquirol Hospital Center, Limoges, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No